CLINICAL TRIAL: NCT01799993
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Safety and Efficacy of BAY 41-6551 as Adjunctive Therapy in Intubated and Mechanically-Ventilated Patients With Gram-Negative Pneumonia
Brief Title: Inhaled Amikacin Solution BAY41-6551 as Adjunctive Therapy in the Treatment of Gram-Negative Pneumonia
Acronym: INHALE 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13084; 2013-001048-73 (EudraCT Number); NCT00805168 (obsolete NCT alias)
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Results first posted 2018-06-26 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Pneumonia, Bacterial
Keywords: Gram-negative pneumonia; Intubation; Mechanical ventilation; Amikacin
MeSH Terms: conditions — Pneumonia, Bacterial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Amikacin inhale (BAY41-6551) (Experimental): Participants received 400 mg (3.2 mL) aerosolized Amikacin (BAY41-6551) solution every 12 hours via Pulmonary Drug Delivery System (PDDS) Clinical from Day 1 to Day 10.
  Interventions: Drug: Amikacin Inhalation Solution (BAY41-6551)
- Placebo (Placebo Comparator): Participants received 3.2 mL aerosolized placebo solution every 12 hours via PDDS Clinical from Day 1 to Day 10.
  Interventions: Drug: Aerosolized Placebo

INTERVENTIONS:
Drug: Amikacin Inhalation Solution (BAY41-6551) — 400 mg of aerosolized amikacin every 12 hours for 10 days to be administered using the Pulmonary Drug Delivery System (PDDS Clinical)
  Arms: Amikacin inhale (BAY41-6551)
Drug: Aerosolized Placebo — Aerosolized placebo every 12 hours for 10 days to be administered using the Pulmonary Drug Delivery System (PDDS Clinical)
  Arms: Placebo

SUMMARY:
To demonstrate that as adjunctive therapy to intravenous (IV) antibiotics, BAY 41-6551 400 mg (amikacin as free base) administered as an aerosol by the Pulmonary Drug Delivery System (PDDS) Clinical every 12 hours is safe and more effective than placebo (aerosolized normal saline) administered as an aerosol by the PDDS Clinical every 12 hours, in intubated and mechanically-ventilated patients with Gram-negative Pneumonia. The secondary endpoint objectives are to evaluate the superiority of aerosolized BAY 41-6551 versus aerosolized placebo in pneumonia-related mortality, the Early Clinical Response at Day 10, the days on ventilation, and the days in the intensive care unit (ICU).

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant, non-lactating females, 18 years of age or older
* Intubated and mechanically-ventilated
* Diagnosis of pneumonia defined as presence of a new or progressive infiltrate(s) on chest radiograph
* Presence of Gram-negative organism(s) by either Gram stain or culture of respiratory secretions, or suspected Gram-negative pathogen
* Impaired oxygenation
* Clinical Pulmonary Infection Score (CPIS) of at least 6
* Presence of a multi-drug resistant (MDR) organism in a pre-therapy respiratory specimen OR at least two risk factors for MDR organisms

Exclusion Criteria:

* History of hypersensitivity to amikacin or other aminoglycosides
* Has received antibiotic therapy for Gram-negative pneumonia for greater than 48 hours at the time of randomization
* Known or suspected bacteremia secondary to Staphylococcus aureus
* A positive urine and/or serum beta-human Chorionic Gonadotropin pregnancy test
* Patients with a serum creatinine > 2 mg/dL (177 µmol/L) [Exception: Patients with a serum creatinine > 2 mg/dL (177 µmol/L) and being treated with continuous renal replacement therapy (Continuous Veno-Venous Hemodialysis and CVVHemoDiafiltration) or daily hemodialysis will receive the aerosol study drug treatment]
* Has been on mechanical ventilation for > 28 days
* Is participating in or has participated in other investigational interventional studies within the last 28 days prior to study treatment
* The risk of rapidly fatal illness and death within 72 hrs, or any concomitant condition not related to ventilator-associated pneumonia that, in the opinion of the investigator, precludes completion of study evaluations and the course of therapy
* Has an Acute Physiology and Chronic Health Evaluation (APACHE) II score < 10
* Patients receiving veno-venous extracorporeal circulation membrane oxygenation (V-V ECMO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 725 (Actual)
Dates: Start 2013-04-13 (Actual); Primary Completion 2017-04-07 (Actual); Study Completion 2017-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (59):
- United States (30):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Phoenix, Arizona
  - Danbury, Connecticut
  - Hartford, Connecticut
  - Newark, Delaware
  - Hollywood, Florida
  - Miami, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Springfield, Illinois
  - Muncie, Indiana
  - Iowa City, Iowa
  - Hazard, Kentucky
  - Kalamazoo, Michigan
  - Springfield, Missouri
  - St Louis, Missouri
  - Butte, Montana
  - Las Vegas, Nevada
  - Brooklyn, New York
  - Mineola, New York
  - New York, New York
  - Asheville, North Carolina
  - Greensboro, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Youngstown, Ohio
  - Oklahoma City, Oklahoma
  - Charleston, South Carolina
- Australia (3):
  - Blacktown, New South Wales
  - Clayton, Victoria
  - Wollongong
- Brazil (3):
  - Belo Horizonte, Minas Gerais
  - Campinas, São Paulo
  - São José do Rio Preto, São Paulo
- Canada (5):
  - Kingston, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec
- Colombia (2):
  - Barranquilla, Atlántico
  - Cali, Valle del Cauca Department
- Czechia (2):
  - Prague
  - Zlín
- Mexico (5):
  - Guadalajara, Jalisco
  - México, D.F., Mexico City
  - Monterrey, Nuevo León
  - Aguascalientes
  - San Luis Potosí City
- Quezon City, Philippines
- Seoul, South Korea
- Taiwan (3):
  - Kaohsiung City
  - Tainan
  - Taipei
- Thailand (2):
  - Chiang Mai
  - Khon Kaen
- Turkey (Türkiye) (2):
  - Ankara
  - Trabzon

REFERENCES:
- [Derived] Niederman MS, Alder J, Bassetti M, Boateng F, Cao B, Corkery K, Dhand R, Kaye KS, Lawatscheck R, McLeroth P, Nicolau DP, Wang C, Wood GC, Wunderink RG, Chastre J. Inhaled amikacin adjunctive to intravenous standard-of-care antibiotics in mechanically ventilated patients with Gram-negative pneumonia (INHALE): a double-blind, randomised, placebo-controlled, phase 3, superiority trial. Lancet Infect Dis. 2020 Mar;20(3):330-340. doi: 10.1016/S1473-3099(19)30574-2. Epub 2019 Dec 19. PMID 31866328
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: To shorten the time required to obtain data from the 2 clinical studies of Amikacin Inhale Phase 3 program, Bayer and the FDA decided that the results of studies NCT01799993 and NCT00805168 should be consolidated into a single report. The studies were conducted at 166 centers across 25 countries, between 13 APR 2013 (FPFV) and 07 APR 2017 (LPLV).
Pre-assignment Details: A total of 807 participants were screened, of which 725 participants were randomized for the 2 studies (264 for NCT01799993 and 461 for NCT00805168), 712 participants were treated with study treatment per exposure data in EDC; 354 received aerosolized amikacin inhale and 358 received placebo.
Period: Overall Study
Arm/Group | Amikacin Inhale (BAY41-6551) | Placebo
Started | 362 | 363
ITT Population | 354 | 358
mITT Population | 255 | 253
Completed (Completed follow-up) | 229 | 235
Not Completed | 133 | 128
Not completed — Didn't complete CRF page "End of FU" | 30 | 40
Not completed — Death | 61 | 45
Not completed — Withdrawal by Subject | 23 | 24
Not completed — Lost to Follow-up | 5 | 8
Not completed — Withdrawal by parent/guardian/LAR | 5 | 3
Not completed — Protocol driven decision point | 0 | 3
Not completed — Protocol Violation | 1 | 1
Not completed — Deterioration of general conditions | 2 | 0
Not completed — Screen failure | 0 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Recovery | 0 | 1
Not completed — Logistical difficulties | 1 | 0
Not completed — Protocol deviation | 1 | 0
Not completed — Non-compliance with medical device | 1 | 0
Not completed — Withdrawal by parent/guardian | 0 | 1
Not completed — Other | 1 | 0
Not completed — Subject didn't return for follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population (included all subjects who were treated with at least one dose of study drug)
Groups:
- Total: Total of all reporting groups
Arm/Group | Amikacin Inhale (BAY41-6551) | Placebo | Total
Number analyzed (Participants) | 354 | 358 | 712
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.8 (15.78) | 64.1 (17.04) | 63.9 (16.42)
Age, Customized [Count of Participants; unit: Participants]
  <18 | 0 | 0 | 0
  18 to <45 | 38 | 53 | 91
  45 to <65 | 130 | 105 | 235
  65 to <75 | 92 | 83 | 175
  >=75 | 94 | 117 | 211
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 107 | 214
  Male | 247 | 251 | 498
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 49 | 55 | 104
  Not Hispanic or Latino | 262 | 250 | 512
  Unknown or Not Reported | 43 | 53 | 96
APACHE II score [Count of Participants; unit: Participants] — The Acute Physiology and Chronic Health Evaluation II (APACHE II) is a severity of disease classification system (Knaus et al, 1985), one of several ICU scoring systems. After admission of a patient to an ICU, an integer score from 0 to 71 is computed based on several measurements; higher scores imply a more severe disease and a higher risk of death. Participants who met all of the inclusion criteria and none of the exclusion criteria were stratified by geographic region (or country) and disease severity using APACHE II score, and randomized in a 1:1 ratio to one of the two treatment groups.
  Participants
    <20 | 187 | 186 | 373
    >=20 | 167 | 172 | 339
CPIS [Mean (Standard Deviation); unit: Scores on a scale] — The Clinical Pulmonary Infection Score (CPIS) is an accepted tool for clinical estimation of ventilator-associated pneumonia (VAP), encompassing five components: tracheal secretions (volume and purulence), temperature, blood leukocytes, oxygenation (P/F ratio). An integer point score from 0 to 2 is assigned for each component; the total CPIS point score (ranges from 0 to 10) is calculated as the sum of the five components ; higher scores imply a more severe disease.
  Scores on a scale | 7.1 (1.38) | 6.9 (1.29) | 7.0 (1.34)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Surviving Through LFU Visit
Description: The primary efficacy variable is Survival through the late follow-up (LFU) visit. Survival is achieved when the participant is alive through the LFU visit. No other factors are considered in the evaluation of survival.
Time Frame: Up to 28-32 days after start of study treatment
Population: Modified intent-to-treat (mITT) population (included all subjects who had a culture-confirmed Gram-negative bacteria that had been treated with at least one dose of study treatment, and had an APACHE II score ≥ 10 at the time of diagnosis of pneumonia)
Measure: Count of Participants; unit: Participants
Arm/Group | Amikacin Inhale (BAY41-6551) | Placebo
Number analyzed (Participants) | 255 | 253
Participants
  Clinical Success (Survive) | 191 | 196
  Clinical Failure (Did not survive) | 64 | 57
Statistical Analysis 1: Comparison: Amikacin Inhale (BAY41-6551) vs Placebo; Test type: Superiority; p = 0.4263, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.841, 95% CI 2-sided [0.554 to 1.277]

2. Secondary Outcome: Number of Participants With Adjudicated Pneumonia-Related Death Through LFU Visit
Description: Death through LFU visit was adjudicated as pneumonia-related or pneumonia-unrelated for participants in the amikacin inhale group and participants in the placebo group.
Time Frame: Up to 28-32 days after start of study treatment
Population: Participants who died through LFU visit in mITT population set
Measure: Count of Participants; unit: Participants
Arm/Group | Amikacin Inhale (BAY41-6551) | Placebo
Number analyzed (Participants) | 64 | 57
Participants
  Pneumonia-related mortality | 43 | 36
  Pneumonia-unrelated mortality | 21 | 21
Statistical Analysis 1: Comparison: Amikacin Inhale (BAY41-6551) vs Placebo; Test type: Superiority; p = 0.6421, Chi-squared

3. Secondary Outcome: Number of Participants With Early Clinical Response
Description: Early Clinical Response was determined by the following: 1. CPIS scoring at Days 3, 5, and 10 compared to baseline (a. On Day 3, CPIS increase from baseline by at least 2 points was considered a failure. b. On Day 5, CPIS decrease from baseline of at least 1 point was not a failure. CPIS of no change from baseline was considered a failure. Any CPIS increase from baseline was a failure. c. On Day 10, CPIS decrease from baseline of at least 2 points was not a failure. CPIS decrease of only 1 point is a failure. Clinical Pulmonary Infection Score of no change was considered a failure. Any CPIS increase from baseline was a failure). 2. All-cause mortality through EOT visit was a failure. 3. The development of empyema or lung abscess through the EOT visit was a failure.
Time Frame: Up to 10 days after start of study treatment
Population: mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Amikacin Inhale (BAY41-6551) | Placebo
Number analyzed (Participants) | 255 | 253
Participants
  Early Clinical Response - Success | 149 | 145
  Early Clinical Response - Failure | 106 | 108
Statistical Analysis 1: Comparison: Amikacin Inhale (BAY41-6551) vs Placebo; Test type: Superiority; p = 0.7984, Chi-squared

4. Secondary Outcome: Number of Days on Mechanical Ventilation Through LFU Visit
Description: Number of days on mechanical ventilator was summarized by descriptive statistics. Duration was defined as the number of days from the date of first study drug through the LFU visit. For participants who lived through the LFU visit, the ventilation days were actual days on ventilation with a maximum value of 28 days. For participants who died after Day 28 but on or before their LFU visit, the days on ventilator was censored at 28 days. For participants who died or discontinued off ventilation, the number of days on ventilation was actual days on ventilation with a maximum value of 28 days. For participants who died or discontinued on ventilation, the number of days on ventilation was 28 days. Further analysis of the number of days on mechanical ventilator was to be performed with censoring at Day 28 for subset of participants on ventilation without censoring.
Time Frame: Up to 28-32 days after start of study treatment
Population: mITT population
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Amikacin Inhale (BAY41-6551) | Placebo
Number analyzed (Participants) | 255 | 253
day | 20.6 (10.09) | 20.2 (10.24)
Statistical Analysis 1: Comparison: Amikacin Inhale (BAY41-6551) vs Placebo; Test type: Superiority; p = 0.7144, ANOVA

5. Secondary Outcome: Number of Days in the ICU Through LFU Visit
Description: Number of days in ICU was summarized by descriptive statistics. Duration was defined as the number of days from the date of first study drug through the LFU visit. For participants who lived in ICU through the LFU visit, the ICU days were actual days in ICU with a maximum value of 28 days. For participants who died after Day 28 but on or before their LFU visit, the days in ICU was censored at 28 days. For participants who died or discontinued in ICU, the number of days in ICU was 28 days. Further analysis of the number of days in ICU was to be performed with censoring at Day 28 for subset of participants on ventilation and without censoring.
Time Frame: Up to 28-32 days after start of study treatment
Population: mITT population without missing start or end dates
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Amikacin Inhale (BAY41-6551) | Placebo
Number analyzed (Participants) | 247 | 249
day | 21.3 (8.17) | 21.9 (7.99)
Statistical Analysis 1: Comparison: Amikacin Inhale (BAY41-6551) vs Placebo; Test type: Superiority; p = 0.4278, ANOVA

6. Other Pre Specified Outcome: Number of Participants With Microbiological Response Per Pathogen at TOC Visit
Description: The number of participants with microbiological response for each pathogen among the total number of participants with baseline pathogen isolates for each pathogen was determined. If a participant had 3 pathogens, all 3 were tabulated. Eradication ( defined as the absence of the original pathogen(s) at the post-treatment test-of-cure [TOC] visit culture of specimens from the original site of infection) and presumed eradication (defined as absence of appropriate culture material in a participant judged to be a clinical cure; he or she was unable to produce sputum and invasive procedures were not warranted) rates were reported to reveal the microbiological responses. The data were displayed for each bacterial genus/species. Baseline pathogen was defined as pathogens tested at Screening and Day 1 visit by central laboratory.
Time Frame: Up to 17-19 days after start of study treatment
Population: mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Amikacin Inhale (BAY41-6551) | Placebo
Number analyzed (Participants) | 255 | 253
Participants
  Achromobacter xylosoxidans: number analyzed (Participants) | 1 | 2
  Achromobacter xylosoxidans | 0 | 2
  Acinetobacter: number analyzed (Participants) | 2 | 0
  Acinetobacter | 1 | 0
  Acinetobacter anitratus: number analyzed (Participants) | 77 | 69
  Acinetobacter anitratus | 46 | 43
  Acinetobacter junii: number analyzed (Participants) | 1 | 0
  Acinetobacter junii | 1 | 0
  Burkholderia cepacia complex: number analyzed (Participants) | 2 | 2
  Burkholderia cepacia complex | 1 | 1
  Chryseobacterium indologenes: number analyzed (Participants) | 0 | 1
  Chryseobacterium indologenes | 0 | 1
  Citrobacter farmeri: number analyzed (Participants) | 1 | 0
  Citrobacter farmeri | 1 | 0
  Citrobacter freundii complex: number analyzed (Participants) | 4 | 6
  Citrobacter freundii complex | 3 | 4
  Citrobacter koseri: number analyzed (Participants) | 7 | 2
  Citrobacter koseri | 3 | 2
  Corynebacterium argentoratense: number analyzed (Participants) | 1 | 0
  Corynebacterium argentoratense | 1 | 0
  Corynebacterium propinquum: number analyzed (Participants) | 0 | 1
  Corynebacterium propinquum | 0 | 0
  Corynebacterium striatum: number analyzed (Participants) | 2 | 1
  Corynebacterium striatum | 2 | 0
  Elizabethkingia meningoceptica: number analyzed (Participants) | 1 | 1
  Elizabethkingia meningoceptica | 1 | 1
  Enterobacter aerogenes: number analyzed (Participants) | 4 | 5
  Enterobacter aerogenes | 4 | 2
  Enterobacter cloacae: number analyzed (Participants) | 15 | 16
  Enterobacter cloacae | 9 | 10
  Enterococcus faecalis: number analyzed (Participants) | 1 | 2
  Enterococcus faecalis | 1 | 2
  Enterococcus faecium: number analyzed (Participants) | 1 | 1
  Enterococcus faecium | 1 | 1
  Escherichia coli: number analyzed (Participants) | 28 | 29
  Escherichia coli | 21 | 19
  Ewingella americana: number analyzed (Participants) | 0 | 1
  Ewingella americana | 0 | 1
  Haemophilus influenzae: number analyzed (Participants) | 10 | 10
  Haemophilus influenzae | 8 | 10
  Haemophilus parahaemolyticus: number analyzed (Participants) | 1 | 0
  Haemophilus parahaemolyticus | 1 | 0
  Haemophilus parainfluenzae: number analyzed (Participants) | 1 | 0
  Haemophilus parainfluenzae | 1 | 0
  Hafnia alvei: number analyzed (Participants) | 2 | 2
  Hafnia alvei | 1 | 2
  Kerstersia gyiorum: number analyzed (Participants) | 1 | 1
  Kerstersia gyiorum | 1 | 0
  Klebsiella oxytoca: number analyzed (Participants) | 3 | 7
  Klebsiella oxytoca | 2 | 5
  Klebsiella pneumoniae: number analyzed (Participants) | 53 | 44
  Klebsiella pneumoniae | 38 | 28
  Kluyvera intermedia: number analyzed (Participants) | 1 | 0
  Kluyvera intermedia | 1 | 0
  Moraxella catarrhalis: number analyzed (Participants) | 1 | 3
  Moraxella catarrhalis | 1 | 3
  Morganella morganii: number analyzed (Participants) | 1 | 0
  Morganella morganii | 0 | 0
  Neisseria: number analyzed (Participants) | 2 | 1
  Neisseria | 2 | 0
  Pantoea agglomerans: number analyzed (Participants) | 1 | 0
  Pantoea agglomerans | 1 | 0
  Pasteurella multocida: number analyzed (Participants) | 1 | 0
  Pasteurella multocida | 1 | 0
  Proteus mirabilis: number analyzed (Participants) | 3 | 10
  Proteus mirabilis | 2 | 6
  Proteus vulgaris: number analyzed (Participants) | 1 | 0
  Proteus vulgaris | 0 | 0
  Providencia stuartii: number analyzed (Participants) | 0 | 1
  Providencia stuartii | 0 | 1
  Pseudomonas aeruginosa: number analyzed (Participants) | 75 | 88
  Pseudomonas aeruginosa | 55 | 44
  Pseudomonas putida: number analyzed (Participants) | 1 | 1
  Pseudomonas putida | 0 | 1
  Raoultella ornithinolytica: number analyzed (Participants) | 1 | 0
  Raoultella ornithinolytica | 0 | 0
  Raoultella planticola: number analyzed (Participants) | 4 | 3
  Raoultella planticola | 3 | 2
  Serratia liquefaciens: number analyzed (Participants) | 1 | 0
  Serratia liquefaciens | 1 | 0
  Serratia marcescens: number analyzed (Participants) | 16 | 17
  Serratia marcescens | 12 | 13
  Staphylococcus aureus: number analyzed (Participants) | 16 | 15
  Staphylococcus aureus | 12 | 10
  Staphylococcus haemolyticus: number analyzed (Participants) | 1 | 0
  Staphylococcus haemolyticus | 1 | 0
  Stenotrophomonas maltophilia: number analyzed (Participants) | 16 | 16
  Stenotrophomonas maltophilia | 12 | 10
  Streptococcus agalactiae: number analyzed (Participants) | 2 | 2
  Streptococcus agalactiae | 2 | 2
  Streptococcus anginosus group: number analyzed (Participants) | 0 | 1
  Streptococcus anginosus group | 0 | 1
  Streptococcus mitis group: number analyzed (Participants) | 4 | 1
  Streptococcus mitis group | 2 | 0
  Streptococcus pneumoniae: number analyzed (Participants) | 2 | 0
  Streptococcus pneumoniae | 2 | 0

7. Other Pre Specified Outcome: Number of Participants With Microbiological Response at TOC Visit
Description: The responses of eradication (defined as the absence of the original pathogen(s) at the post-treatment TOC culture of specimens from the original site of infection) and presumed eradication (defined as absence of appropriate culture material in a participant judged to be a clinical cure; he or she was unable to produce sputum and invasive procedures were not warranted) were tabulated for each participant to reveal the microbiological responses. All pathogen isolates from a participant must be eradicated (or presumed eradicated) to tabulate an eradicated (or presumed eradicated) response. Baseline pathogen was defined as pathogens tested at Screening and Day 1 visit by central laboratory.
Time Frame: Up to 17-19 days after start of study treatment
Population: mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Amikacin Inhale (BAY41-6551) | Placebo
Number analyzed (Participants) | 255 | 253
Participants | 150 | 118

8. Other Pre Specified Outcome: Number of Participants With Microbiological Recurrence at LFU Visit
Description: The responses of recurrence were tabulated for each participant. Recurrence was defined as the reappearance of the original pathogen(s) from a specimen taken after the TOC visit. If one or more pathogen reappeared, all isolates from a participant were tabulated as "recurrence". Baseline pathogen was defined as pathogens tested at Screening and Day 1 visit by central laboratory.
Time Frame: Up to 28-32 days after start of study treatment
Population: mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Amikacin Inhale (BAY41-6551) | Placebo
Number analyzed (Participants) | 255 | 253
Participants | 12 | 12

9. Other Pre Specified Outcome: Number of Participants With Emergence of New Respiratory Pathogens During the Aerosol Treatment Period
Description: New pathogens also denoted as superinfection was defined as the isolation of a new pathogen (not the original baseline pathogen) from a specimen taken while the participant was on antibiotic therapy (Day 1 to EOT) and having a need for alternative antimicrobial therapy. Rates of emergence of any new pathogen by participant after start of study drug were summarized for each treatment group.
Time Frame: Up to 10 days after start of study treatment
Population: mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Amikacin Inhale (BAY41-6551) | Placebo
Number analyzed (Participants) | 255 | 253
Participants | 21 | 34

10. Other Pre Specified Outcome: Number of Participants With Emergence of Resistance Among Pathogens
Description: Resistance to amikacin was determined for the bacterial isolates by using a standardized microbiology laboratory test that generates a minimum inhibitory concentration (MIC) for amikacin and bacterial isolate. The same microbiology resistance standard was used for all bacteria tested against amikacin. Resistant bacteria have a MIC value of 64 μg/mL or greater. Percentages of resistance were calculated based on the percentage of participants infected with any treatment-emergent pathogens resistant to amikacin. If a participant had a more than one occurrence of a specific pathogen during pre-treatment period, the worst case of testing was used.
Time Frame: Up to 28-32 days after start of study treatment
Population: mITT population participants with pathogen susceptible to amikacin in pre-treatment period
Measure: Count of Participants; unit: Participants
Arm/Group | Amikacin Inhale (BAY41-6551) | Placebo
Number analyzed (Participants) | 186 | 194
Participants | 13 | 17

11. Other Pre Specified Outcome: Number of Participants Who Received at Least One Dose of Study Drug and Reported an Adverse Event
Description: AE was untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. AEs, occurred any time after the first dose of therapy and through 7 days after the EOT were recorded as treat-emergent AEs (TEAEs).
Time Frame: Up to 7 days after the end of study treatment
Population: ITT for Safety population (included all participants in ITT analysis set who were analyzed as treated for safety analyses)
Measure: Count of Participants; unit: Participants
Arm/Group | Amikacin Inhale (BAY41-6551) | Placebo
Number analyzed (Participants) | 353 | 359
Participants | 295 | 303

12. Other Pre Specified Outcome: Number of Participants Who Received at Least One Dose of Study Drug and Reported a Serious Adverse Event
Description: AE was untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. Serious AE: AE resulting in following outcomes or deemed significant for any reason: death; life-threatening; inpatient hospitalization or prolongation of existing hospitalization; persistent; significant disability/incapacity; congenital anomaly/birth defect; medical important serious event judged by investigator. SAEs, occurred any time after the first dose of therapy and through 7 days after the EOT were recorded as treat-emergent SAEs (TESAEs).
Time Frame: Up to 7 days after the end of study treatment
Population: ITT for Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Amikacin Inhale (BAY41-6551) | Placebo
Number analyzed (Participants) | 353 | 359
Participants | 101 | 97

13. Other Pre Specified Outcome: Number of Participants With Organ Failure
Description: The overall number of participants with any organ failure was summarized for each treatment group. Organ failure was defined by a specific organ type and by a collection of MedDRA version 20.0 preferred terms that were determined by the sponsor's clinical team. A participant with multiple AEs within a system organ class or preferred term is counted a single time for that system organ class (SOC) or preferred term.
Time Frame: Up to 7 days after the end of study treatment
Population: ITT for Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Amikacin Inhale (BAY41-6551) | Placebo
Number analyzed (Participants) | 353 | 359
Participants | 69 | 67

14. Other Pre Specified Outcome: Number of Death Due to Any Reason Through Day 10 and Day 15
Description: Number of deaths due to any reason through Day 10 and Day 15 were summarized for each treatment group.
Time Frame: Up to 10 days and 15 days after start of study treatment, respectively
Population: mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Amikacin Inhale (BAY41-6551) | Placebo
Number analyzed (Participants) | 255 | 253
Participants
  Number of death through Day 10 | 23 | 32
  Number of death through Day 15 | 32 | 39

ADVERSE EVENTS:
Time Frame: After the first dose of study drug and no later than 7 days after end of treatment
Groups:
- Amikacin Inhale 400mg q12h: Patients received 400 mg (3.2 mL) aerosolized Amikacin (BAY41-6551) solution every 12 hours via PDDS Clinical from Day 1 to Day 10.
- Placebo: Patients received 3.2 mL placebo solution aerosolized every 12 hours via PDDS Clinical from Day 1 to Day 10.
Arm/Group | Amikacin Inhale 400mg q12h | Placebo
All-Cause Mortality (participants affected / at risk) | 86/353 | 85/359
Serious Adverse Events (participants affected / at risk) | 101/353 | 97/359
Other Adverse Events (participants affected / at risk) | 207/353 | 214/359
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amikacin Inhale 400mg q12h (N=353) | Placebo (N=359)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (3) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 5 (5) | 3 (3)
Cardiac failure (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 3 (3) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 5 (5) | 5 (5)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 3 (3) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Mediastinitis (Infections and infestations) | 1 (1) | 0 (0)
Pathogen resistance (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 5 (5)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 5 (5) | 4 (4)
Septic shock (Infections and infestations) | 7 (7) | 15 (15)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 1 (1)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1)
Bacillus bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Brain herniation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumonitis chemical (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Weaning failure (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Respiratory rate decreased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain hypoxia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Stroke in evolution (Nervous system disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 4 (4)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 4 (5)
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Reexpansion pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 3 (3) | 2 (2)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (2)
Device malfunction (Product Issues) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amikacin Inhale 400mg q12h (N=353) | Placebo (N=359)
Anaemia (Blood and lymphatic system disorders) | 36 (38) | 44 (49)
Coagulopathy (Blood and lymphatic system disorders) | 5 (5) | 10 (11)
Atrial fibrillation (Cardiac disorders) | 9 (9) | 10 (10)
Tachycardia (Cardiac disorders) | 6 (6) | 11 (11)
Constipation (Gastrointestinal disorders) | 30 (30) | 32 (32)
Diarrhoea (Gastrointestinal disorders) | 27 (30) | 33 (34)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 13 (13) | 6 (6)
Vomiting (Gastrointestinal disorders) | 6 (7) | 17 (18)
Oedema (General disorders) | 5 (5) | 9 (9)
Oedema peripheral (General disorders) | 9 (12) | 13 (14)
Pyrexia (General disorders) | 18 (21) | 21 (24)
Hepatic function abnormal (Hepatobiliary disorders) | 12 (12) | 13 (13)
Septic shock (Infections and infestations) | 8 (11) | 5 (5)
Urinary tract infection (Infections and infestations) | 10 (11) | 10 (10)
Oxygen saturation decreased (Investigations) | 5 (5) | 8 (10)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (8) | 10 (11)
Hyperkalaemia (Metabolism and nutrition disorders) | 14 (14) | 10 (10)
Hypernatraemia (Metabolism and nutrition disorders) | 9 (9) | 12 (12)
Hypoglycaemia (Metabolism and nutrition disorders) | 5 (5) | 9 (12)
Hypokalaemia (Metabolism and nutrition disorders) | 32 (36) | 37 (40)
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 (9) | 7 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 17 (17) | 12 (12)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (6) | 11 (11)
Hypoproteinaemia (Metabolism and nutrition disorders) | 8 (9) | 4 (4)
Metabolic alkalosis (Metabolism and nutrition disorders) | 8 (10) | 10 (10)
Agitation (Psychiatric disorders) | 8 (8) | 12 (12)
Delirium (Psychiatric disorders) | 14 (15) | 9 (9)
Insomnia (Psychiatric disorders) | 6 (6) | 11 (11)
Oliguria (Renal and urinary disorders) | 3 (3) | 8 (8)
Renal impairment (Renal and urinary disorders) | 4 (4) | 9 (9)
Acute kidney injury (Renal and urinary disorders) | 9 (9) | 7 (9)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 10 (15) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 9 (9)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 11 (11) | 14 (14)
Hypertension (Vascular disorders) | 13 (13) | 7 (8)
Hypotension (Vascular disorders) | 23 (24) | 12 (12)
Deep vein thrombosis (Vascular disorders) | 9 (9) | 3 (3)

LIMITATIONS AND CAVEATS:
To shorten the time required to obtain data from the 2 clinical studies of Amikacin Inhale Phase 3 program, Bayer and the FDA decided that the results of studies NCT01799993 and NCT00805168 should be consolidated into a single report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI will not make any publication of the results of the Study before the first multi-center publication, unless otherwise agreed upon by the Parties. In the event there is no multi-center publication within eighteen (18) months after a Study has been completed or terminated as all Study sites, Institution and/or Investigator shall have the right to publish the results from the Study at the Institution subject to the guideline laid out in the contacts.

DOCUMENTS (2):
  • Study Protocol (2017-08-29): https://cdn.clinicaltrials.gov/large-docs/93/NCT01799993/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT01799993/SAP_001.pdf